CLINICAL TRIAL: NCT00602680
Title: A Multicenter, Double-blind, Parallel-group, Placebo-controlled Study of the Effect on Cognitive Performance and Safety/Tolerability of SSR180711C for 4 Weeks, Using Donepezil as Calibrator, in Patients With Mild Alzheimer's Disease
Brief Title: Effect on Cognitive Performance and Safety/Tolerability of SSR180711C in Mild Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient expected benefit risk
Sponsor: Sanofi (Industry)
Responsible Party: ICD study director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PDY10400; SSR180711; EudraCT 2007-001639-80
Record Dates: First submitted 2008-01-16; First posted 2008-01-28 (Estimated); Last update posted 2009-07-20 (Estimated); Status verified 2009-07

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer; cognitive
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental): dose 1
  Interventions: Drug: SSR180711C
- 2 (Experimental): dose 2
  Interventions: Drug: SSR180711C
- 3 (Experimental): dose 3
  Interventions: Drug: SSR180711C
- 4 (Placebo Comparator)
  Interventions: Drug: placebo
- 5 (Active Comparator)
  Interventions: Drug: donepezil

INTERVENTIONS:
Drug: SSR180711C — duration of treatment: 4 weeks
  Arms: 1; 2; 3
Drug: donepezil — duration of treatment: 4 weeks
  Arms: 5
Drug: placebo — duration of treatment: 4 weeks
  Arms: 4

SUMMARY:
The primary objective of the study is to assess the effect of 3 doses of SSR180711C on cognitive performance in patients with mild Alzheimer's Disease (AD). Other objectives are to assess the safety/tolerability of SSR180711C in patients with mild AD.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with diagnosis of mild AD

Exclusion Criteria:

* Concomitant or previous treatment by acetylcholinesterase inhibitors and/or memantine
* Medical condition which may interfere with the study
* History of epileptic seizures
* Lens opacity
* Lack of reliable caregiver

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Change in cognitive performance | 4 weeks

SECONDARY OUTCOMES:
Cognitive, global, functional and behaviorial assessments | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bruno DUBOIS, MD, Study Chair — Scientific Advisory Committee
Locations (1):
- Sanofi-Aventis Administrative Office, Paris, France